CLINICAL TRIAL: NCT02903368
Title: Phase II Randomized Study Of Neoadjuvant And Adjuvant Abiraterone Acetate + Apalutamide For Intermediate-High Risk Prostate Cancer Undergoing Prostatectomy
Brief Title: Neoadjuvant And Adjuvant Abiraterone Acetate + Apalutamide Prostate Cancer Undergoing Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Mary-Ellen Taplin, MD, Mary-Ellen Taplin, MD, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-223
Record Dates: First submitted 2016-08-24; First posted 2016-09-16 (Estimated); Results first posted 2021-09-05 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: abiraterone acetate; apalutamide; leuprolide; prednisone; neoadjuvant therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Leuprolide; luprolide acetate gel depot; Prednisone; Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1A: AAPL Neoadjuvant Therapy [Part 1] (Experimental): Eligible Participants will be randomized to receive:
  AAPL: Abiraterone acetate (240 mg/day orally), Apalutamide (1000 mg/day orally), Leuprolide (22.5 mg every 12 weeks intramuscularly), Prednisone (5 mg/twice daily orally) for 6 months
  Pts x weeks to RP
  Interventions: Drug: Apalutamide; Drug: Leuprolide; Drug: Prednisone; Drug: Abiraterone Acetate
- Arm 1B: APL Neoadjuvant Therapy [Part 1] (Experimental): Eligible Participants will be randomized to receive:
  APL: Abiraterone acetate (1000 mg/day orally), Leuprolide (22.5 mg every 12 weeks intramuscularly), Prednisone (5 mg/day orally) for 6 months
  Interventions: Drug: Leuprolide; Drug: Prednisone; Drug: Abiraterone Acetate
- Arm 2A: AAPL Adjuvant Therapy [Part 2] (Experimental): Eligible Participants will be randomized to receive:
  AAPL: Abiraterone acetate (240 mg/day orally), Apalutamide (1000 mg/day orally), Leuprolide (22.5 mg every 12 weeks intramuscularly), Prednisone (5 mg/twice daily orally) for 12 months
  Interventions: Drug: Apalutamide; Drug: Leuprolide; Drug: Prednisone; Drug: Abiraterone Acetate
- Arm 2B: Observation [Part 2] (No Intervention)

INTERVENTIONS:
Drug: Apalutamide
  Other Names: JNJ-56021927; ARN-509
  Arms: Arm 1A: AAPL Neoadjuvant Therapy [Part 1]; Arm 2A: AAPL Adjuvant Therapy [Part 2]
Drug: Leuprolide
  Other Names: Lupron; Eligard
  Arms: Arm 1A: AAPL Neoadjuvant Therapy [Part 1]; Arm 1B: APL Neoadjuvant Therapy [Part 1]; Arm 2A: AAPL Adjuvant Therapy [Part 2]
Drug: Prednisone
  Other Names: Deltasone
  Arms: Arm 1A: AAPL Neoadjuvant Therapy [Part 1]; Arm 1B: APL Neoadjuvant Therapy [Part 1]; Arm 2A: AAPL Adjuvant Therapy [Part 2]
Drug: Abiraterone Acetate
  Other Names: Zytiga
  Arms: Arm 1A: AAPL Neoadjuvant Therapy [Part 1]; Arm 1B: APL Neoadjuvant Therapy [Part 1]; Arm 2A: AAPL Adjuvant Therapy [Part 2]

SUMMARY:
This multicenter randomized phase II trial investigates the impact of intense androgen deprivation on radical prostatectomy (RP) pathologic response and radiographic and tissue biomarkers in localized prostate cancer (NCT02903368).

DETAILED DESCRIPTION:
This is a multicenter, phase II, prospective, randomized trial designed to investigate the efficacy of neoadjuvant and adjuvant abiraterone acetate + apalutamide for men with intermediate-high risk prostate cancer who are candidates for RP.

The study includes two parts. In part 1, patients will be randomized in 1:1 ratio to receive 6 months of abiraterone acetate, apalutamide, leuprolide and prednisone (Arm 1A) versus 6 months of abiraterone acetate, leuprolide and prednisone (Arm 1B) followed by RP, stratified by risk factor (intermediate versus high-risk). High-risk factors will be defined as a Gleason score ≥ 8, PSA > 20 ng/dL, or T3 disease on MRI.

In part 2 (post-RP), patients will be randomized in 1:1 ratio to receive an additional 12 months of abiraterone acetate, apalutamide, leuprolide and prednisone (Arm 2A) or observation (Arm 2B) stratified by type of neoadjuvant therapy and pathological T-stage (< pT3 versus ≥ pT3) after RP but before cycle 7 day 1 following neoadjuvant therapy. There will be an early stopping rule for Part 2 should a high rate of patients refuse to participate or drop out early while receiving adjuvant therapy (<6 months).

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥ 18 years of age.
2. Histologically confirmed adenocarcinoma of the prostate without histological variants comprising >50% of the sample as determined by academic center central review (including neuroendocrine differentiation, small cell, sarcomatoid, ductal adenocarcinoma, squamous or transitional cell carcinoma).
3. Must have 3 core biopsies involved with cancer (a minimum of 6 core biopsies must be obtained). Prostate biopsy must be within seven months from screening. Less than 3 core biopsies are allowed if the patient has >1 cm or T3 disease on MRI.
4. Patients must have the following features:

   * Gleason ≥ 4+3=7 OR
   * Gleason 3+4=7 AND at least one of the following: PSA >20 ng/dL or T3 disease (as determined by MRI).
5. No evidence of metastatic disease as determined by radionuclide bone scans and CT/MRI. Lymph nodes must be less than 20 mm in the short (transverse) axis.
6. Participants must be candidates for RP and considered surgically resectable by urologic evaluation.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
8. Participants must have normal organ and marrow function as defined below:

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1,500/mcL
   * Platelets ≥ 100,000/mcL, independent of transfusions/growth factors within 3 months of treatment start
   * Serum potassium ≥ 3.5 mmol/L
   * Serum total bilirubin ≤ 2.0 x upper limit of normal (ULN) (except in subjects with Gilbert's syndrome who have a total bilirubin > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤ 1.5 x ULN, subject may be eligible)
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN
   * Serum albumin ≥ 3.0 g/dL
   * Serum creatinine < 2.0 x ULN
   * PTT≤60
9. Participant must agree to use a condom (even men with vasectomies) and another effective method of birth control if having sex with a woman of childbearing potential or must agree to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Participant must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug.
10. Medications known to lower the seizure threshold (see list under APPENDIX D: Representative Medications that May Predispose to Seizure) must be discontinued or substituted at least 1 week prior to study treatment.

Exclusion Criteria:

1. Prior hormone therapy for prostate cancer including orchiectomy, antiandrogens (including first-generation antiandrogens, enzalutamide, Apalutamide and others), CYP17 inhibitors (including abiraterone acetate, TAK-700, galeterone, ketoconazole, and others), estrogens, Luteinizing Hormone Releasing Hormone (LHRH) agonist/antagonists. Prior therapy with 5α-reductase inhibitors is allowed. LHRH therapy allowed if begun within 4 weeks of day 1.
2. Prior chemotherapy, radiation therapy, or immunotherapy for prostate cancer.
3. Prior systemic treatment with an azole drug within two weeks of start of treatment.
4. Hypogonadism or severe androgen deficiency as defined by screening serum testosterone < 200 ng/dL.
5. Clinically significant cardiovascular disease within 6 months of study treatment including:

   * Severe or unstable angina;
   * Myocardial infarction;
   * Symptomatic congestive heart failure;
   * New York Heart Association (NYHA) class II-IV heart disease;
   * Arterial or venous thromboembolic events (such as pulmonary embolism cerebrovascular accident including transient ischemic attacks);
   * History of clinically significant ventricular arrhythmias (e.g. ventricular tachycardia, ventricular fibrillation, torsades de pointes);
   * Prolonged corrected QT interval by the Fridericia correction formula (QTcF) on screening EKG > 470 msec;
   * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place;
   * Uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg). Participants with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive therapy.
6. History of seizure or any condition or concurrent medication that may predispose to seizure (including but not limited to prior stroke, transient ischemic attack, loss of consciousness within 1 year prior to randomization, brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect).
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Apalutamide, abiraterone acetate, or other study drugs.
8. Severe hepatic impairment (Child-Pugh Class C).
9. Active infection (such as human immunodeficiency virus (HIV) or viral hepatitis) or other medical condition that would make prednisone / prednisolone corticosteroid use contraindicated.
10. History of pituitary or adrenal dysfunction.
11. Gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug.
12. Pre-existing condition that warrants long-term corticosteroid use greater than the equivalent of 10 mg prednisone daily. Physiologic replacement is permitted. Topical, intra-articular, or inhaled corticosteroids are permitted.
13. Concomitant use of medications that may alter pharmacokinetics of abiraterone acetate or Apalutamide.
14. Individuals with a history of a different malignancy are ineligible except for the following circumstances: 1) individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy, or 2) individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: non-muscle invasive bladder cancer, basal cell or squamous cell carcinoma of the skin.
15. Major surgery or radiation therapy within 30 days of screening visit. Participants who have had a major surgery within 30 days of screening visit may be eligible provided the treating investigator deems that the participant is at low risk for complications.
16. Any condition that in the opinion of the investigator would preclude participation in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2024-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - University of California, San Diego Moores Cancer Center, La Jolla, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McKay RR, Xie W, Yang X, Acosta A, Rathkopf D, Laudone VP, Bubley GJ, Einstein DJ, Chang P, Wagner AA, Kane CJ, Preston MA, Kilbridge K, Chang SL, Choudhury AD, Pomerantz MM, Trinh QD, Kibel AS, Taplin ME. Postradical prostatectomy prostate-specific antigen outcomes after 6 versus 18 months of perioperative androgen-deprivation therapy in men with localized, unfavorable intermediate-risk or high-risk prostate cancer: Results of part 2 of a randomized phase 2 trial. Cancer. 2024 May 1;130(9):1629-1641. doi: 10.1002/cncr.35170. Epub 2024 Jan 1. PMID 38161319
- [Derived] McKay RR, Xie W, Ye H, Fennessy FM, Zhang Z, Lis R, Calagua C, Rathkopf D, Laudone VP, Bubley GJ, Einstein DJ, Chang PK, Wagner AA, Parsons JK, Preston MA, Kilbridge K, Chang SL, Choudhury AD, Pomerantz MM, Trinh QD, Kibel AS, Taplin ME. Results of a Randomized Phase II Trial of Intense Androgen Deprivation Therapy prior to Radical Prostatectomy in Men with High-Risk Localized Prostate Cancer. J Urol. 2021 Jul;206(1):80-87. doi: 10.1097/JU.0000000000001702. Epub 2021 Mar 8. PMID 33683939

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a 2-part study:
  In part 1, patients will be randomized in 1:1 ratio to receive 6 months of AAPL (Arm 1A) versus 6 months of APL (Arm 1B) followed by RP, stratified by risk factor.
  In part 2 (post-RP), patients will be randomized in 1:1 ratio to receive an additional 12 months of AAPL (Arm 2A) or observation (Arm 2B) stratified by type of neoadjuvant therapy and pathological T-stage after RP but before cycle 7 day 1 following neoadjuvant therapy.
Pre-assignment Details: The part 2 of the study is still in progression and the final data has not been collected
Groups:
- Arm 1A: AAPL Neoadjuvant Therapy (Part 1): Eligible participants will be randomized to receive:
  AAPL: Abiraterone acetate (240 mg/day orally), Apalutamide (1000 mg/day orally), Leuprolide (22.5 mg every 12 weeks intramuscularly), Prednisone (5 mg/twice daily orally) for 6 months.
- Arm 1B: APL Neoadjuvant Therapy (Part 1): Eligible Participants will be randomized to receive:
  APL: Abiraterone acetate (1000 mg/day orally), Leuprolide (22.5 mg every 12 weeks intramuscularly), Prednisone (5 mg/day orally) for 6 months
- Arm 2A: AAPL Adjuvant Therapy (Part 2): Eligible participants will be randomized to receive adjuvant AAPL post surgery: Abiraterone acetate (240 mg/day orally), Apalutamide (1000 mg/day orally), Leuprolide (22.5 mg every 12 weeks intramuscularly), Prednisone (5 mg/twice daily orally) for 12 months
- Arm 2B: Observation (Part 2): Eligible participants will be randomized to the observation arm post surgery
Period: Part 1
Arm/Group | Arm 1A: AAPL Neoadjuvant Therapy (Part 1) | Arm 1B: APL Neoadjuvant Therapy (Part 1) | Arm 2A: AAPL Adjuvant Therapy (Part 2) | Arm 2B: Observation (Part 2)
Started | 59 | 59 | 0 | 0
Completed | 55 | 59 | 0 | 0
Not Completed | 4 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Part 2
Arm/Group | Arm 1A: AAPL Neoadjuvant Therapy (Part 1) | Arm 1B: APL Neoadjuvant Therapy (Part 1) | Arm 2A: AAPL Adjuvant Therapy (Part 2) | Arm 2B: Observation (Part 2)
Started (Only 82 patients underwent part 2 randomization; the remaining 36 patients did not participate in part 2 randomization.) | 0 | 0 | 42 | 40
Completed | 0 | 0 | 31 | 38
Not Completed | 0 | 0 | 11 | 2
Not completed — Adverse Event | 0 | 0 | 5 | 0
Not completed — Subject withdrew after 6 cycles of protocol therapy. | 0 | 0 | 1 | 0
Not completed — Subject withdrew after part-2 randomization and remained on observation. | 0 | 0 | 4 | 0
Not completed — Subject withdrew after part-2 randomization and received non-protocol therapy. | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1A: AAPL Neoadjuvant Therapy (Part 1) | Arm 1B: APL Neoadjuvant Therapy (Part 1) | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Continuous [Median (Full Range); unit: years] | 62 [47 to 72] | 58 [46 to 72] | 61 [46 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 59 | 59 | 118
Race/Ethnicity, Customized [Number; unit: participants]
  White | 55 | 48 | 103
  Black or African American | 3 | 6 | 9
  Asian | 0 | 2 | 2
  Other | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 59 | 59 | 118

OUTCOME MEASURES:

1. Primary Outcome: Combined pCR or MRD Rate [Part 1]
Description: Pathological response, defined as achieving either pCR or MRD at radical prostatectomy (RP). Pathological Complete Response (pCR) is defined as the absence of morphologically identifiable carcinoma in the RP specimen. MRD will be defined as residual tumor in the RP specimen measuring ≤ 5 mm.
Time Frame: Assessed from RP specimens, at 6 months from the initiation of neoadjuvant therapy.
Population: 114 patients (55 in AAPL Arm and 59 in APL Arm) had RP pathologic assessment, excluding the four who withdrew prior to RP.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A: AAPL Neoadjuvant Therapy (Part 1) | Arm 1B: APL Neoadjuvant Therapy (Part 1)
Number analyzed (Participants) | 55 | 59
Participants | 12 | 12

2. Primary Outcome: Biochemical Progression Free Survival (bPFS) Rate at 3 Years Post RP [Part 2]
Description: 3-year bPFS rate is defined as the probability of biochemical progression free and survival at 3 years from the date of Part 2 randomization, which is estimated using Kaplan Meier methods. The event is considered to be biochemical progression (defined as a confirmed PSA ≥ 0.2 ng/mL), local, regional, or distant metastatic disease on CT/MRI or bone scan, or receipt of post-operative systemic therapy or radiotherapy for rising PSA, or death from any cause. Participants who are lost to follow-up before the 3-year mark are censored at date last disease evaluation.
Time Frame: At 3 years post RP
Population: The primary efficacy analysis was the intent-to-treat approach, including all patients who have been randomized into Part 2 of the study.
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Arm/Group | Arm 2A: AAPL Adjuvant Therapy (Part 2) | Arm 2B: Observation (Part 2)
Number analyzed (Participants) | 42 | 40
percentage of subjects | 81 [68 to 89] | 72 [59 to 82]

3. Secondary Outcome: Rate of pCR at RP (Part 1)
Description: Pathological Complete Response (pCR) is defined as the absence of morphologically identifiable carcinoma in the RP specimen at radical prostatectomy (RP).
Time Frame: Assessed from RP specimens, at 6 months from the initiation of neoadjuvant therapy.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A: AAPL Neoadjuvant Therapy (Part 1) | Arm 1B: APL Neoadjuvant Therapy (Part 1)
Number analyzed (Participants) | 55 | 59
Participants | 7 | 6

4. Secondary Outcome: Median of Residual Cancer Burden (RCB) at RP (Part 1)
Description: RCB was calculated as "tumor volume (cm^3) X % cellularity". RCB was analyzed as a continuous score (with median and range) instead of a categorical variable based on the percentile cutoff point, at the time of radical prostatectomy (RP).
Time Frame: Assessed from RP specimens, at 6 months from the initiation of neoadjuvant therapy.
Population: as for outcome 1
Measure: Median (Full Range); unit: (cm^3) * %
Arm/Group | Arm 1A: AAPL Neoadjuvant Therapy (Part 1) | Arm 1B: APL Neoadjuvant Therapy (Part 1)
Number analyzed (Participants) | 55 | 59
(cm^3) * % | 0.023 [0 to 7.8] | 0.075 [0 to 6.8]

5. Secondary Outcome: Frequency of Presenting Cribriform at RP (Part 1)
Description: Presence or cribriform was evaluated by central pathology review of specimens at radical prostatectomy (RP).
Time Frame: Assessed from RP specimens, at 6 months from the initiation of neoadjuvant therapy.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A: AAPL Neoadjuvant Therapy (Part 1) | Arm 1B: APL Neoadjuvant Therapy (Part 1)
Number analyzed (Participants) | 55 | 59
Participants | 1 | 0

6. Secondary Outcome: Frequency of Presenting Intraductal Carcinoma at RP (Part 1)
Description: Intraductal carcinoma was evaluated by central pathology review of specimens at Radical Prostatectomy (RP).
Time Frame: Assessed from RP specimens, at 6 months from the initiation of neoadjuvant therapy.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A: AAPL Neoadjuvant Therapy (Part 1) | Arm 1B: APL Neoadjuvant Therapy (Part 1)
Number analyzed (Participants) | 55 | 59
Participants | 15 | 19

7. Secondary Outcome: Frequency of Positive Surgical Margins at RP (Part 1)
Description: Pathologic specimens were centrally reviewed and counted for positive surgical margins at the time of Radical Prostatectomy (RP).
Time Frame: Assessed from RP specimens, at 6 months from the initiation of neoadjuvant therapy.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A: AAPL Neoadjuvant Therapy (Part 1) | Arm 1B: APL Neoadjuvant Therapy (Part 1)
Number analyzed (Participants) | 55 | 59
Participants | 4 | 7

8. Secondary Outcome: Percent of Participants With Nadir PSA < 0.2 ng/mL Prior to RP (Part 1)
Description: Prostate specific antigen (PSA) was measured on day 1 of each cycle during the neoadjuvant therapy. PSA nadir was defined as the lowest PSA value prior to Radical Prostatectomy (RP). Number and percent of participants with nadir PSA < 0.2 ng/mL were reported.
Time Frame: Assessed on day 1 of each cycle (1 cycle=28 +/- 2 days), up to 6 months from the initiation of neoadjuvant therapy.
Population: PSA nadir was collected in 115 patients (56 in AAPL Arm and 59 in APL Arm).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A: AAPL Neoadjuvant Therapy (Part 1) | Arm 1B: APL Neoadjuvant Therapy (Part 1)
Number analyzed (Participants) | 56 | 59
Participants | 55 | 58

9. Secondary Outcome: Frequency of Presenting Intra-operative Complications Following RP (Part 1)
Description: Intra-operative complications were collected via questionnaire following Radical Prostatectomy.
Time Frame: Assessed post-RP, at 6 months from the initiation of neoadjuvant therapy.
Population: Assessed in 114 patients (55 in AAPL Arm and 59 in APL Arm) who received RP, excluding the four who withdrew prior to RP.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A: AAPL Neoadjuvant Therapy (Part 1) | Arm 1B: APL Neoadjuvant Therapy (Part 1)
Number analyzed (Participants) | 55 | 59
Participants | 1 | 1

10. Secondary Outcome: Biochemical Progression Free Survival (bPFS) Rate at 2 Years Post RP [Part 2]
Description: 2-year bPFS rate is defined as the probability of biochemical progression free and survival at 2 years from the date of Part 2 randomization, which is estimated using Kaplan Meier methods. The event is considered to be biochemical progression (defined as a confirmed PSA ≥ 0.2 ng/mL), local, regional, or distant metastatic disease on CT/MRI or bone scan, or receipt of post-operative systemic therapy or radiotherapy for rising PSA, or death from any cause. Participants who are lost to follow-up before the 2-year mark are censored at date of last disease evaluation.
Time Frame: At 2 years post RP
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Arm/Group | Arm 2A: AAPL Adjuvant Therapy (Part 2) | Arm 2B: Observation (Part 2)
Number analyzed (Participants) | 42 | 40
percentage of subjects | 90 [79 to 96] | 80 [67 to 88]

11. Secondary Outcome: Biochemical Progression Free Survival (bPFS) Rate at 4 Years Post RP [Part 2]
Description: 4-year bPFS rate is defined as the probability of biochemical progression free and survival at 4 years from the date of Part 2 randomization, which is estimated using Kaplan Meier methods. The event is considered to be biochemical progression (defined as a confirmed PSA ≥ 0.2 ng/mL), local, regional, or distant metastatic disease on CT/MRI or bone scan, or receipt of post-operative systemic therapy or radiotherapy for rising PSA, or death from any cause. Participants who are lost to follow-up before the 4-year mark are censored at date of last disease evaluation.
Time Frame: At 4 years post RP
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Arm/Group | Arm 2A: AAPL Adjuvant Therapy (Part 2) | Arm 2B: Observation (Part 2)
Number analyzed (Participants) | 42 | 40
percentage of subjects | 67 [53 to 78] | 61 [47 to 73]

12. Secondary Outcome: Rate of Freedom From Further Anti-cancer Therapy at 2-years Post RP (Part 2)
Description: Defined as the probability of freedom from further anti-cancer therapy at 2-years from the date of Part 2 randomization, which is estimated using Kaplan Meier methods. The event includes initiation of anti-cancer therapy (radiation therapy, ADT, or other therapies) for rising PSAs and/or clinical progression. Participants who are lost to follow-up before the 2-year mark are censored at date of last follow-up.
Time Frame: At 2-years post RP
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Arm/Group | Arm 2A: AAPL Adjuvant Therapy (Part 2) | Arm 2B: Observation (Part 2)
Number analyzed (Participants) | 42 | 40
percentage of subjects | 90 [80 to 96] | 80 [67 to 88]

13. Secondary Outcome: Rate of Freedom From Further Anti-cancer Therapy at 3-years Post RP (Part 2)
Description: Defined as the probability of freedom from further anti-cancer therapy at 3-years from the date of Part 2 randomization, which is estimated using Kaplan Meier methods. The event includes initiation of anti-cancer therapy (radiation therapy, ADT, or other therapies) for rising PSAs and/or clinical progression. Participants who are lost to follow-up before the 3-year mark are censored at date of last follow-up.
Time Frame: At 3 years post RP
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Arm/Group | Arm 2A: AAPL Adjuvant Therapy (Part 2) | Arm 2B: Observation (Part 2)
Number analyzed (Participants) | 42 | 40
percentage of subjects | 83 [71 to 91] | 72 [59 to 82]

14. Secondary Outcome: Rate of Freedom From Further Anti-cancer Therapy at 4-years Post RP (Part 2)
Description: Defined as the probability of freedom from further anti-cancer therapy at 4-years from the date of Part 2 randomization, which is estimated using Kaplan Meier methods. The event includes initiation of anti-cancer therapy (radiation therapy, ADT, or other therapies) for rising PSAs and/or clinical progression. Participants who are lost to follow-up before the 4-year mark are censored at date of last follow-up.
Time Frame: At 4-years post RP
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Arm/Group | Arm 2A: AAPL Adjuvant Therapy (Part 2) | Arm 2B: Observation (Part 2)
Number analyzed (Participants) | 42 | 40
percentage of subjects | 78 [65 to 87] | 67 [53 to 78]

15. Secondary Outcome: Mean Scores for Quality of Life (QOL) Questionnaires EPIC-26 at 6-months Post-RP (Part 2)
Description: The QOL will be measured using the Expanded Prostate Cancer Index Composite 26 (EPIC-26). For part 2, the questionnaires will be administered at 6 months, 12 months, and 24 months post RP. Resulting domain scores for EPIC-26 (urinary incontinence, urinary obstruction, sexual, bowel, hormonal/vitality) is on a 0-100 scale, with higher values representing a more favorable health-related QOL.
Time Frame: At 6-months post-RP
Population: 32 subjects receiving Arm 2A and 34 receiving Arm 2B completed EPIC-26 QOL questionnaires at 6 months post RP.
Measure: Mean (Standard Deviation); unit: Score on 0-100
Arm/Group | Arm 2A: AAPL Adjuvant Therapy (Part 2) | Arm 2B: Observation (Part 2)
Number analyzed (Participants) | 32 | 34
Score on 0-100
  Urinary Irritative | 90 (11) | 92 (8)
  Urinary Incontinence | 63 (24) | 72 (23)
  Bowel | 95 (11) | 96 (7)
  Sexual | 17 (19) | 14 (14)
  Hormonal | 68 (20) | 83 (16)

16. Secondary Outcome: Mean Scores for Quality of Life (QOL) Questionnaires EPIC-26 at 12-months Post-RP (Part 2)
Description: as for outcome 15
Time Frame: At 12-months post-RP
Population: 32 subjects receiving Arm 2A and 39 receiving Arm 2B completed EPIC-26 QOL questionnaires at 12 months post RP.
Measure: Mean (Standard Deviation); unit: score on 0-100 scale
Arm/Group | Arm 2A: AAPL Adjuvant Therapy (Part 2) | Arm 2B: Observation (Part 2)
Number analyzed (Participants) | 32 | 39
score on 0-100 scale
  Urinary Irritative | 91 (11) | 91 (10)
  Urinary Incontinence | 75 (24) | 74 (25)
  Bowel | 95 (12) | 94 (12)
  Sexual | 16 (18) | 26 (26)
  Hormonal | 68 (22) | 86 (15)

17. Secondary Outcome: Mean Scores for Quality of Life (QOL) Questionnaires EPIC-26 at 24-months Post-RP (Part 2)
Description: as for outcome 15
Time Frame: At 24-months post-RP
Population: 14 subjects receiving Arm 2A and 12 receiving Arm 2B completed EPIC-26 QOL questionnaires at 24 months post RP. The QOL questionnaire completion rate was low at the 24-month visit. Due to the Covid19 pandemic, many follow-up visits were conducted virtually. These questionnaires were done when possible and the patients were back in the clinic.
Measure: Mean (Standard Deviation); unit: score on 0-100 scale
Arm/Group | Arm 2A: AAPL Adjuvant Therapy (Part 2) | Arm 2B: Observation (Part 2)
Number analyzed (Participants) | 14 | 12
score on 0-100 scale
  Urinary Irritative | 92 (12) | 93 (9)
  Urinary Incontinence | 75 (22) | 76 (30)
  Bowel | 95 (12) | 97 (4)
  Sexual | 31 (31) | 26 (30)
  Hormonal | 88 (20) | 90 (8)

ADVERSE EVENTS:
Time Frame: Part 1: Adverse events (AE) and Serious AEs (SAE) during neoadjuvant therapy collected on Day 1 of each cycle (+/-2 days) from the first dose of the study drugs until 30 days after discontinuation of the neoadjuvant therapy, up to 7 months from treatment initiation. Part 2: AE and SAE during adjuvant therapy collected from the date informed consent is signed (for Part 2) until 30 days after discontinuation from adjuvant treatment, up to 13 months from adjuvant treatment initiation.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Groups:
- Arm 2A: AAPL Adjuvant Therapy (Part 2): Eligible participants will be randomized to receive adjuvant AAPL post surgery: Abiraterone acetate (240 mg/day orally), Apalutamide (1000 mg/day orally), Leuprolide (22.5 mg every 12 weeks intramuscularly), Prednisone (5 mg/twice daily orally) for 12 months
  Of the 42 patients randomized to Arm 2A, only 37 patients received the AAPL treatment; 5 patients declined protocol treatment after part-2 randomization. Therefore, toxicities for Arm 2A were reported among the 37 patients who actually received AAPL treatment.
- Arm 2B: Observation (Part 2): Eligible participants will be randomized to the observation arm post surgery.
  Of the 40 patients randomized to Arm 2B (observation), 38 remained on observation and 2 received non-protocol therapy. Therefore, the AE analysis for Arm 2B included the 38 patients on observation, excluding 2 patient receiving non-protocol therapy.
Arm/Group | Arm 1A: AAPL Neoadjuvant Therapy (Part 1) | Arm 1B: APL Neoadjuvant Therapy (Part 1) | Arm 2A: AAPL Adjuvant Therapy (Part 2) | Arm 2B: Observation (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59 | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 8/59 | 5/59 | 4/37 | 0/38
Other Adverse Events (participants affected / at risk) | 59/59 | 59/59 | 30/37 | 28/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1A: AAPL Neoadjuvant Therapy (Part 1) (N=59) | Arm 1B: APL Neoadjuvant Therapy (Part 1) (N=59) | Arm 2A: AAPL Adjuvant Therapy (Part 2) (N=37) | Arm 2B: Observation (Part 2) (N=38)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 5 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1A: AAPL Neoadjuvant Therapy (Part 1) (N=59) | Arm 1B: APL Neoadjuvant Therapy (Part 1) (N=59) | Arm 2A: AAPL Adjuvant Therapy (Part 2) (N=37) | Arm 2B: Observation (Part 2) (N=38)
Abdominal infection (Infections and infestations) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Agitation (Psychiatric disorders) | 2 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 14 | 22 | 1 | 1
Alkaline phosphatase increased (Investigations) | 0 | 2 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 4 | 8 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 13 | 20 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 5 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Cholesterol high (Investigations) | 4 | 3 | 3 | 2
Cognitive disturbance (Nervous system disorders) | 2 | 1 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 3 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 3 | 0
Creatinine increased (Investigations) | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 2 | 4 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 4 | 1
Dizziness (Nervous system disorders) | 3 | 4 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 1
Dysgeusia (Nervous system disorders) | 5 | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dysphasia (Nervous system disorders) | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 0
Edema limbs (General disorders) | 2 | 1 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 10 | 13 | 0 | 2
Facial pain (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 30 | 30 | 10 | 1
Fever (General disorders) | 0 | 2 | 0 | 1
Flashing lights (Eye disorders) | 1 | 0 | 0 | 0
Flu like symptoms (General disorders) | 1 | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 4 | 2 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Gynecomastia (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Headache (Nervous system disorders) | 8 | 11 | 3 | 1
Hematuria (Renal and urinary disorders) | 1 | 3 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 | 2 | 0 | 0
Hot flashes (Vascular disorders) | 51 | 50 | 2 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Hypertension (Vascular disorders) | 16 | 11 | 10 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 1 | 0 | 1
Injection site reaction (General disorders) | 2 | 1 | 0 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 9 | 6 | 0 | 1
Investigations - Other, specify (Investigations) | 1 | 1 | 1 | 0
Irritability (General disorders) | 1 | 1 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Libido decreased (Psychiatric disorders) | 3 | 7 | 0 | 0
Localized edema (General disorders) | 0 | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 2 | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 5 | 8 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 6 | 2 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 4 | 2 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 3 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Personality change (Psychiatric disorders) | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0
Pleural infection (Infections and infestations) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 | 3 | 3 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3 | 1 | 0 | 0
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 | 0 | 0 | 3
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1
Skin infection (Infections and infestations) | 0 | 0 | 2 | 0
Small intestinal mucositis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0
Testicular disorder (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 0
Urethral anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 7 | 6 | 3 | 0
Urinary incontinence (Renal and urinary disorders) | 22 | 21 | 4 | 8
Urinary retention (Renal and urinary disorders) | 2 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 3 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1 | 0
Weight gain (Investigations) | 1 | 3 | 1 | 2
Weight loss (Investigations) | 0 | 2 | 1 | 0
White blood cell decreased (Investigations) | 0 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT02903368/Prot_SAP_000.pdf